CLINICAL TRIAL: NCT06172218
Title: Prospective, Randomized Controlled Pilot Study Assessing Micronized Amniotic Membrane and Umbilical Cord Particulate in Patients With Symptomatic and Refractory Achilles Tendinopathy
Brief Title: AM for Refractory Achilles Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: North Park Podiatry (Other)
Responsible Party: Principal Investigator, Trent Brookshier, Podiatrist/ Founder, North Park Podiatry
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-001
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Achilles Tendinopathy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micronized Amniotic Membrane (Experimental): Injection of micronized amniotic membrane reconstituted in 2.0 mL sterile, preservative free 0.9% NaCl
  Interventions: Other: Flo; Other: Saline
- Preservative Free Normal Saline (Placebo Comparator): 2.0 mL sterile, preservative free 0.9% NaCl
  Interventions: Other: Saline

INTERVENTIONS:
Other: Flo — sterile, micronized human amniotic membrane product derived from placenta and umbilical cord
  Arms: Micronized Amniotic Membrane
Other: Saline — sterile, preservative free 0.9% NaCl

SUMMARY:
To evaluate outcomes after use of micronized amniotic membrane to replace or supplement damaged or inadequate integumental tissue in patients with "chronic" insertional or non-insertional Achilles tendinopathy that remains refractory to standard care. Outcomes between a control and treatment group in this pilot study will be used to devise a multi-center study with larger sample size.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 64 years old
2. BMI ≤ 40 kg/m2
3. Subject has been diagnosed with unilateral Achilles tendinopathy (based on investigator assessment using ultrasound) of at least 3 months duration
4. History of having attempted a physical therapy for Achilles tendinopathy which must have included at least 6 weeks of eccentric exercise, alone or in addition to other non-surgical therapies
5. VISA-A score for the target tendon ≥40 and ≤60 at screening
6. Subject is willing to comply with all study procedures
7. Willing to sign a written informed consent to participate
8. Able to follow study instructions, with the intention of completing all required visits

Exclusion Criteria:

1. Planned surgical procedure below knee of the targeted extremity during study period
2. Patient has previously received an injection for this injury within the past 2 months
3. Major lower limb amputation of the contralateral leg
4. A medical condition, or a personal situation, which in the principal investigator's opinion, is not appropriate for participation in the trial
5. Osteoarthritis, chronic low back pain, fibromyalgia or any other condition that may affect the responses on the VISA-A
6. HIV infection, Hepatitis B or C infection, tuberculosis, COVID-19, cellulitis or any other active infection
7. Cognitive impairment, mental illness, neuroses, or untreated depression that would preclude understanding or reliably completing the patient reported outcome measures
8. Peritendinopathy, paratenonitis, partial tear or tendon rupture of the affected tendon
9. Subject has hindfoot deformities on the targeted extremity
10. Plantar fasciitis, calcaneal bursitis, Sever's disease, retrocalcaneal exostosis (Mulholland deformity, Haglund's deformity), enthesophytes, myofascial pain referral, posterior ankle impingement, os trigonum syndrome, tenosynovitis or dislocation of the peroneal or other plantar flexor tendons, an accessory soleus muscle, irritation or neuroma of the sural nerve, or systemic inflammatory disease
11. Leg length discrepancy, hyperpronation, varus deformity of the forefoot, pes cavus or limited mobility of the subtalar joint
12. Prior surgical intervention to the affected tendon
13. Current use of vitamins or herbal supplements
14. Current use of opioids, midazolam, gabapentin, pregabalin or ketamine
15. Compensable disability or work injury, ongoing litigation, or ongoing chiropractic care
16. Current use of systemic immunosuppressive medications, chemotherapy, or history of organ transplant (kidney, heart, lung)
17. Pregnancy and women who are expecting to be pregnant
18. Current enrollment in another interventional drug or device study or participation in such a study within 30 days of anticipated entry into this study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-04-28 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
Change in Achilles pain | 30 days
  A score of 0 is considered no pain while a score of 10 is considered very severe pain

SECONDARY OUTCOMES:
Change from Baseline in NRS score | over 3 months
  A score of 0 is considered no pain while a score of 10 is considered very severe pain
Change from Baseline in VISA-A score | over 3 months
Proportion of responders based on change in VISA-A score | over 3 months
  20 points as a threshold for assignment of responder status
Proportion of complete pain relief | over 3 months
  pain score of 0
Time to complete pain relief | over 3 months
  pain score of 0
Proportion of subjects that respond feeling at least better and satisfied | 3 months
  patient satisfaction survey

CONTACTS AND LOCATIONS:
Locations (1):
- North Park Podiatry, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided